CLINICAL TRIAL: NCT02372006
Title: Phase I/II Open Label, Dose Escalation Trial to Determine the MTD, Safety, PK and Efficacy of Afatinib Monotherapy in Children Aged ≥1 Year to <18 Years With Recurrent/Refractory Neuroectodermal Tumours, Rhabdomyosarcoma and/or Other Solid Tumours With Known ErbB Pathway Deregulation Regardless of Tumour Histology
Brief Title: Trial of Afatinib in Pediatric Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.120; 2014-002123-10 (EudraCT Number)
Record Dates: First submitted 2015-02-24; First posted 2015-02-26 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Neuroectodermal Tumors; Rhabdomyosarcoma
MeSH Terms: conditions — Neuroectodermal Tumors; Rhabdomyosarcoma | interventions — Afatinib

ARMS (1):
- afatinib (Experimental): dose escalation
  Interventions: Drug: afatinib

INTERVENTIONS:
Drug: afatinib

SUMMARY:
Open-label, dose escalation, monotherapy, basket trial with biomarker specific MTD expansion cohort/Phase II part.

The trial will consist of 2 parts:

1. Dose finding part to determine the MTD
2. Biomarker specific MTD expansion cohort/Phase II part to assess clinical anti-tumour activity in included tumour types

ELIGIBILITY:
Inclusion criteria:

* Paediatric patients aged 1 year to <18 years at the time of informed consent
* diagnosis of HGG, DIPG, low grade astrocytoma, medulloblastoma/PNET, ependymoma, neuroblastoma, RMS and tumours with ErbB deregulation
* recurrent/refractory disease after they received at least one prior standard treatment regimen
* no effective conventional therapy exists
* Performance status >= 50% (Lansky for =<12ys; Karnofsky for >12ys)
* Further inclusion criteria apply

Exclusion criteria:

* relevant toxicity from previous treatment
* known pre-existing relevant cardiac , hepatic, renal, bone marrow dysfunction, ILD, keratitis
* Further exclusion criteria apply

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (28):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Sydney Childrens Hospital, Randwick, New South Wales, Australia
- Austria (2):
  - AKH - Medical University of Vienna, Vienna
  - St. Anna Children-Hospital, Children's Cancer Research, Wien, Vienna
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Rigshospitalet, København, Børneonkologisk Afsnit 5002, København Ø, Denmark
- HOP Toulouse, Pédiat, Toulouse, Toulouse, Faroe Islands
- France (5):
  - HOP Pellegrin, Bordeaux
  - CTR Oscar Lambret, Lille
  - CTR Leon Berard, Lyon
  - INS Curie, Paris
  - INS Gustave Roussy, Villejuif
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Essen AöR, Essen
  - Universitätsklinikum Tübingen, Tübingen
- Italy (4):
  - Istituto G. Gaslini, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Osp. Pediatrico Bambin Gesù, Roma
- Erasmus MC - Sophia Kinderziekenhuis, Rotterdam, Netherlands
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid
- United Kingdom (4):
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Geoerger B, Marshall LV, Nysom K, Makin G, Bouffet E, Defachelles AS, Amoroso L, Aerts I, Leblond P, Barahona P, Van-Vlerken K, Fu E, Solca F, Lorence RM, Ziegler DS. Afatinib in paediatric patients with recurrent/refractory ErbB-dysregulated tumours: Results of a phase I/expansion trial. Eur J Cancer. 2023 Jul;188:8-19. doi: 10.1016/j.ejca.2023.04.007. Epub 2023 Apr 20. PMID 37178647
- [Derived] Andrade RC, Boroni M, Amazonas MK, Vargas FR. New drug candidates for osteosarcoma: Drug repurposing based on gene expression signature. Comput Biol Med. 2021 Jul;134:104470. doi: 10.1016/j.compbiomed.2021.104470. Epub 2021 May 7. PMID 34004576
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I/II open label, dose escalation trial to determine the Maximum tolerated dose (MTD), safety, Pharmacokinetics (PK) and efficacy of afatinib monotherapy in children aged ≥1 year to <18 years with recurrent/refractory neuroectodermal tumours, rhabdomyosarcoma and/or other solid tumours with known ErbB pathway deregulation regardless of tumour histology.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Groups:
- Dose Finding - Level 0; Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0: Afatinib, dose level 0. (Once daily at 80% of the recommended adult dose per m2 body surface area [BSA] using allometric scaling):
  Oral solid single-unit film-coated tablets for pediatric patients who are able to swallow them. Oral liquid formulation for patients who cannot swallow the film-coated tablets, or for doses which cannot be achieved by the film-coated tablets, or for pediatric patients who did not accept the film-coated tablets.
  Therapy with afatinib continued as long as the individual patient benefited from the therapy, did not develop secondary malignancy, and did not meet one of the criteria requiring withdrawal from treatment.
  Afatinib in film-coated tablet form can be given in tablets of 20, 30, 40 and 50 mg. The dose in film-coated tablets is related to the free base equivalent to afatinib. The dose of afatinib as capsule and solvent for oral solution is given as a 200 mg capsule to be dissolved in aqueous solvent (2 capsules per 100 milliliter solvent) i.e. 4 milligram per milliliter.
- Dose Finding - Level 1: Afatinib, dose level 1. (Once daily at 100% of the recommended adult dose per m2 body surface area [BSA] using allometric scaling):
  Oral solid single-unit film-coated tablets for pediatric patients who are able to swallow them. Oral liquid formulation for patients who cannot swallow the film-coated tablets, or for doses which cannot be achieved by the film-coated tablets, or for pediatric patients who did not accept the film-coated tablets.
  Therapy with afatinib continued as long as the individual patient benefited from the therapy, did not develop secondary malignancy, and did not meet one of the criteria requiring withdrawal from treatment.
  Afatinib in film-coated tablet form can be given in tablets of 20, 30, 40 and 50 mg. The dose in film-coated tablets is related to the free base equivalent to afatinib. The dose of afatinib as capsule and solvent for oral solution is given as a 200 mg capsule to be dissolved in aqueous solvent (2 capsules per 100 milliliter solvent) i.e. 4 milligram per milliliter.
Period: Overall Study
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Started | 8 | 9 | 39
Completed | 0 | 0 | 0
Not Completed | 8 | 9 | 39
Not completed — Progressive disease | 8 | 7 | 34
Not completed — Dose limiting toxicity | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Other reason for not completing | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) This patient set included all patients enrolled in the trial who were documented to have taken at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0 | Total
Number analyzed (Participants) | 8 | 9 | 39 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.75 (4.83) | 10.44 (5.29) | 10.92 (4.44) | 10.68 (4.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 16 | 24
  Male | 4 | 5 | 23 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 37 | 46
  Unknown or Not Reported | 4 | 4 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 4 | 29 | 36
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 5 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response - Maximum Tolerated Dose Expansion (MTD) Cohort
Description: Number of participants with objective response for maximum tolerated dose expansion (MTD) cohort was reported. The objective response was defined as a best overall response of complete response or partial response based on investigator's assessment according to the institutional response evaluation criteria for the given tumour type, assessed every 8 weeks until progression.
Time Frame: Assessed every 8 weeks until progression of disease, up to 336 days.
Population: Treated set (TS): This patient set included all patients enrolled in the trial who were documented to have taken at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 39
Participants | 3

2. Primary Outcome: Area Under the Curve Over Dosing Interval τ at Steady State (AUCτ,ss) - Dose Finding Part
Description: Area under the curve over dosing interval τ at steady state (AUCτ,ss) for Dose finding part was reported.
Time Frame: Pre-dose before afatinib administration then 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h and 24 h after administration at steady state on Day 8.
Population: Pharmacokinetics (PK) analysis set (PKS): This patient set included all patients in the TS who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with non-missing results were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanogram per milliliter
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1
Number analyzed (Participants) | 7 | 6
hours times nanogram per milliliter | 681 (43.8) | 1380 (29.0)

3. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State (Cmax,ss) - Dose Finding Part
Description: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) for Dose finding part was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1
Number analyzed (Participants) | 7 | 6
nanogram per mililiter | 53.0 (48.8) | 115 (39.3)

4. Primary Outcome: Number of Participants With Dose Limiting Toxicity Adverse Events - Dose Finding Part
Description: Number of participants with Dose Limiting Toxicity adverse events for Dose finding part was reported.
Time Frame: During the first course (28 days) of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1
Number analyzed (Participants) | 8 | 9
Participants | 1 | 2

5. Secondary Outcome: Number of Participants With Objective Response - Dose Finding Part
Description: Number of participants with objective response for Dose finding part was reported. The objective response was defined as a best overall response of complete response or partial response based on investigator's assessment according to the institutional response evaluation criteria for the given tumour type, assessed every 8 weeks until progression.
Time Frame: Assessed every 8 weeks until progression of disease, up to 336 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

6. Secondary Outcome: Progression Free Survival - Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Progression free survival for the MTD expansion cohorts was reported. Progression free survival (PFS) was defined as the duration from the date of first treatment until the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of last adequate tumour assessment.
Time Frame: From the first treatment until date of first progression or death, up to 336 days.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 39
Months | 8.0 [6.4 to 8.29]

7. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to 24 Hours (AUC0-24) - Dose Finding Part
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours (AUC0-24) for Dose finding part was reported.
Time Frame: Pre-dose before afatinib administration then 1 hour (h), 2 h, 3 h, 4 h, 5 h, 6 h, 8 h and 24 h after administration on Day 1.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanogram per mililiter
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1
Number analyzed (Participants) | 8 | 8
hours times nanogram per mililiter | 383 (46.4) | 512 (40.6)

8. Secondary Outcome: Maximum Measured Concentration (Cmax) - Dose Finding Part/Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Maximum measured concentration (Cmax) for Dose finding part/maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 8 | 8 | 36
nanogram per mililiter | 36.4 (55.9) | 43.8 (61.2) | 30.5 (90.3)

9. Secondary Outcome: Time From (Last) Dosing to the Maximum Measured Concentration (Tmax) - Dose Finding Part/Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Time from (last) dosing to the maximum measured concentration (tmax) for Dose finding part/maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 8 | 8 | 36
Hours | 3.02 [2.00 to 6.00] | 3.43 [2.00 to 6.02] | 3.98 [1.00 to 8.00]

10. Secondary Outcome: Time From (Last) Dosing to the Maximum Measured Concentration at Steady State (Tmax,ss) - Dose Finding Part/Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Time from (last) dosing to the maximum measured concentration at steady state (tmax,ss) for Dose finding part/maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 7 | 6 | 25
Hours | 3.00 [2.00 to 6.00] | 2.75 [2.00 to 5.05] | 4.17 [2.00 to 8.00]

11. Secondary Outcome: Accumulation (or Effective) Half-life - Dose Finding Part/Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Accumulation (or effective) half-life for Dose finding part/maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 7 | 6 | 24
hours | 18.7 (44.3) | 31.0 (56.7) | 30.3 (83.6)

12. Secondary Outcome: Duration of Objective Response - Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Duration of objective response in maximum tolerated dose expansion (MTD) cohort was reported. The objective response was defined as a best overall response of complete response or partial response based on investigator's assessment according to the institutional response evaluation criteria for the given tumour type, assessed every 8 weeks until progression.
Time Frame: From first documented response until the earliest of disease progression or death, up to 336 days.
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 39
Days | 62 [57 to 170]

13. Secondary Outcome: Area Under the Curve Over Dosing Interval τ at Steady State (AUCτ,ss) - Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Area under the curve over dosing interval τ at steady state (AUCτ,ss) in maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanogram per milliliter
Arm/Group | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 25
hours times nanogram per milliliter | 780 (60.7)

14. Secondary Outcome: Maximum Measured Concentration of the Analyte in Plasma at Steady State (Cmax,ss) - Maximum Tolerated Dose (MTD) Expansion Cohort
Description: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) in maximum tolerated dose (MTD) expansion cohort was reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter
Arm/Group | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
Number analyzed (Participants) | 25
nanogram per mililiter | 52.5 (61.0)

ADVERSE EVENTS:
Time Frame: From the first drug administration until end of study, up to 336 days.
Description: Treated set (TS) This patient set included all patients enrolled in the trial who were documented to have taken at least one dose of study medication.
Arm/Group | Dose Finding - Level 0 | Dose Finding - Level 1 | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0
All-Cause Mortality (participants affected / at risk) | 8/8 | 9/9 | 29/39
Serious Adverse Events (participants affected / at risk) | 7/8 | 6/9 | 20/39
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Finding - Level 0 (N=8) | Dose Finding - Level 1 (N=9) | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0 (N=39)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2
General physical health deterioration (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Finding - Level 0 (N=8) | Dose Finding - Level 1 (N=9) | Maximum Tolerated Dose (MTD) Expansion Cohort - Level 0 (N=39)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 7
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 3 | 0 | 3
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 2 | 6
Constipation (Gastrointestinal disorders) | 6 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 30
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 15
Oral pain (Gastrointestinal disorders) | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 9
Tongue eruption (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6 | 16
Asthenia (General disorders) | 1 | 0 | 2
Disease progression (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 10
Mucosal inflammation (General disorders) | 0 | 1 | 7
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 5
Xerosis (General disorders) | 0 | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 3
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2
Paronychia (Infections and infestations) | 1 | 0 | 9
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2
Tinea capitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 3 | 4
Neutrophil count decreased (Investigations) | 1 | 0 | 2
Platelet count decreased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 3 | 10
White blood cell count decreased (Investigations) | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 3 | 9
Lethargy (Nervous system disorders) | 0 | 0 | 2
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
VIth nerve disorder (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 9
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 10
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT02372006/SAP_000.pdf
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT02372006/Prot_001.pdf